CLINICAL TRIAL: NCT04289168
Title: Infant Peer Interaction Study by Examining the Effect of a 6-week Music Enhancement Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: research institute on addictions (Unknown)
Responsible Party: Principal Investigator, Kai Ling Kong, Assistant Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Infant PIS
Record Dates: First submitted 2020-02-18; First posted 2020-02-28 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Body Weight Changes
MeSH Terms: conditions — Body Weight Changes | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Class (Experimental): Music Class attendance
  Interventions: Behavioral: Music
- Play Class (No Intervention): Play date class attendance

INTERVENTIONS:
Behavioral: Music — Music class was provided for the intervention group
  Arms: Music Class

SUMMARY:
The overall purpose of this study is to better understand food reinforcement in infants. The results of this study should help to further our understanding of how individuals relate to food and how an enriched environment can change this behavior.

DETAILED DESCRIPTION:
The study will be a between subject design with a Music Together intervention group and a play date active control group. All subjects will complete the orientation and pre-screening intervention assessment sessions.

All infant-mother dyads in the Music together group will attend a 6 weekly, 45-minute classes as a group. Infant-mother dyads will also receive an illustrated songbook with family activities to practice and enjoy at home along with the CD. The program provides CD with a collection of songs, rhythm chants, "play-alongs", tonal and rhythm patterns, which will be used in classes.

All infant-mother dyads in the play date control group will attend 6 weekly, 45-minute organized play dates as a group. These play dates will be planned and led by DBM research staff members. Variety of age-appropriate toys (i.e. puzzles, shape sorters, books) will be provided for the play date. Each family in the play date group will receive a toy from us to practice and play at home with their baby.

Families in both groups are asked to report their home practice with the song or toy with their babies by filling out the Daily Home Practice Survey.

Both groups will attend a post-intervention training assessment session at the conclusion of the 6 week intervention period.

1. Initial email or phone screen:

   Upon receiving an inquiry from a prospective participant, the study will be explained. If the prospective participant has an infant age 9 to 15 months, and she is interested in joining the study, a verbal consent will be obtained in order to screen for eligibility criteria. The initial screening questionnaire could be done via phone or online via Survey Monkey (see Initial Phone Screen/Survey Monkey Questionnaire for details). The information assessed during the initial screen is recorded in a secure database that requires a password. The database is used by select members of the Division of Behavioral Medicine and has been approved for use by previous IRB committees.
2. Orientation:

   If families meet the initial criteria gathered from the initial screen, qualified families will be scheduled for an orientation. At the orientation, there will be an overview of the study. If interested, parents will be asked to review and sign consent forms. Two copies of the consent forms will be signed by all parties involved, person obtaining consent, and the participating parent. One copy will be obtained by the study personnel and one copy will be given to the participants for their records. The copy obtained by study personnel will be kept in a locked cabinet. After signing the consent form, the height and weight of the mother and infant will be measured. She will also be sent a list of links of questionnaires to be completed at home before the further screening/pre-intervention assessment. These questionnaires include the Demographic Questionnaire, Pregnancy History and Infant Feeding Practice Questionnaire, Food Security Questionnaire, Infant Behavior Questionnaires-Revised (IBQ-R), and Baby Eating Behavior Questionnaire (BEBQ). Lastly, before dyads leave, the parent will be asked to list three of their child's favorite foods and rank them on a 7 point Likert type scale anchored by "Do not Like" to "Like very much". Mother will then be asked to provide the child's highest ranked favorite food for the further screening/pre-intervention assessment visit.
3. Further Screening/Pre-Intervention Assessment:

   After orientation, eligible participants will be scheduled for a 45 minute further screening/pre-intervention assessment session. For this visit, the mother will be advised to choose a time of the day when the infant is generally alert, active and ready to play. The infant needs to be fed one hour prior to the lab visit. The mother will be reminded to bring diapers or change of clothes for the infant. The mother will also be reminded not to feed her infant the test food (infant's favorite food) 24 hours before the laboratory visit.

   Then, the mother and infant will be escorted to a laboratory room where the food reinforcement game will take place. Infant will be securely fastened on a high chair. The mother will be in the room with the infant at all-time during the game. The mother will be reminded that the entire reinforcement task procedure will be video recorded to obtain vocalization, body movement and facial expression of the infant. The baseline state of the infant will be assessed. There are five states: 1 = drowsy, 2 = alert/calm, 3 = alert/active, 4 = fussy, 5 = crying. Before the start of the game, a study staff member will go through a training session with the infant to familiarize him/her with the computer based game and button/monitor interface. Mother will be asked to assist with the training by repeating phrases the researchers use during the game. After the training, the study staff member will start the actual game followed by infant's anthropometric measurements.

   After completing all measures, families will be further assessed for eligibility criteria. Eligible participants will be randomly assigned to one of two groups; Music Together program treatment group or the play date control group. Potential participants who are not eligible for the study will be compensated for their time and effort to attend the orientation and further screening/pre-intervention assessment.
4. Intervention The 6-week music intervention, the Music Together® program, was designed in collaboration with a local music studio, Betty's Music Together. This program introduced infants to the pleasures of music making with their parents rather than passively receiving it from CDs or TV. This program provided a rich variety of music and playful activities, which encouraged infants and parents to participate at their own level in singing, moving, listening, or exploring musical instruments. Participating parents and infants attended weekly, 45-minute classes as a group on 6 consecutive Saturday mornings. Besides attending classes, parents were encouraged to listen and sing together with their infants at home during everyday home activities such as bath time, meal time and bed time using the CD and instructional song book provided by the program.

   The active control group consisted of a weekly, 45-minute play date held on the same 6 consecutive Saturday mornings as the music group. Investigators provided a variety of age appropriate toys (no musical toys) and books for participating parents and infants to play with and enjoy. Families in the play date group received a toy, Baby's First Blocks (Fisher-Price®, East Aurora, NY), to practice and play at home.

   Parents in both groups were advised to attend all classes, with an opportunity to attend one makeup session. To encourage families to listen to the Music Together® songs or to play with the Baby's First Blocks daily, investigators sent each family a text reminder every morning Sunday through Friday for the duration of the intervention. Investigators also sent an email Sunday through Friday evenings to remind them to fill out the daily home practice survey. Families that filled out at least five of the daily home practice surveys and attended that week class or play date were entered into a drawing for a $5 gift card to a local grocery or coffee shop.
5. Post-intervention Assessment:

The post-treatment appointment will follow the same structure and timing as the pre-treatment session with the same measurements. Upon completion of all the measures, families will sign their payment form and receive a debriefing sheet.

Further Screening/Pre-Intervention Assessment:

After the orientation, if participant is eligible investigators will schedule a 30 minute visit of further screening/pre-intervention assessment session with participant where participant's baby will perform the second part of the reinforcing game.

Intervention:

After this assessment, if infant-mother dyads are eligible infant-mother dyads will be randomly assigned to Music Together or play date group.

1. Music Together group This program provides CD with a collection of songs, rhythm chants, "play-alongs", tonal and rhythm patterns, which will be used in classes. All infant-mother dyads will attend this 6 weekly, 45-minute classes as a group. Participants will also receive illustrated songbook with family activities to practice and enjoy at home along with the CD.
2. Play date group These play dates will be planned and led by DBM research staff members, which all infant-mother dyads will attend 6 weekly, 45-minute organized play dates as a group. Variety of age-appropriate toys (i.e. puzzles, shape sorters, books) will be provided for the play date. Participants will also receive a toy from us that participants will take home and use to practice and play with participant's baby.

During the six-week intervention, participants will be asked to fill out a Daily Home Practice Survey each day for six days of the week (not on the day participant come for the group meeting).

Post-Intervention Assessment:

At the end of the 6 week intervention infant-mother dyads will come back into the lab for a post-test assessment (2 visits). Infant-mother dyads' height and weight will be measured and payment will be given.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* single birth
* between 9-18 months
* not allergic to puffed grains or cheerios

Exclusion Criteria:

* Your child was premature/preterm at birth (< 37 weeks of gestation)
* Your child had a low birth weight (<2500 grams)
* Your child had any medical problems at birth
* Your child showed signs of developmental delay based on his/her developmental milestones recorded when he/she was 6 to 9 months old
* Infant who are currently participating or previously participated in Music Together® program or similar music program
* Maternal age was less than 18 years at the time of your child's birth
* Mother smoked, used controlled substances (i.e. opiates, cocaine, marijuana) or consumed excessive alcohol during pregnancy
* Mother had a high-risk pregnancy
* Infant who could not complete a food/social interaction reward task during the further screening/pre-intervention assessment
* Your child is not overweight

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 49 (Actual)
Dates: Start 2014-08-11 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
The primary study outcome is the food reinforcing ratio (FRR) | through study completion, an average 13 months
  Infant completed the pre- and post-intervention's FRR task in the lab

SECONDARY OUTCOMES:
Infant weight | through study completion, an average 13 months
  Infant weight were collected pre- and post-intervention in kg
Infant height | through study completion, on average 13 months
  Infant height were collected pre- and post-intervention in cm
Infant zWFL | through study completion, on average 13 months
  Infant zWFL were calculated pre- and post-intervention using the WHO growth chart

CONTACTS AND LOCATIONS:
Overall Officials: Kai ling Kong, Principal Investigator — Assistant Professor